CLINICAL TRIAL: NCT04389684
Title: Clinical and Psycho-Social Impact on Patients With Digestive Tumors of Treatment and Care Modifications Linked to COVID-19 in France
Brief Title: Clinical and Psycho-social Impact of COVID-19 Related Confinement on Patients With Digestive Tumors
Acronym: COVIDICA
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A01301-38
Record Dates: First submitted 2020-05-14; First posted 2020-05-15 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Chemeotherapy; Immunotherapy; Treatment Mofidied; Coronavirus; Quality of Life
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Psycho-Social Questionnaire — Patients, after enrollmenet in the study, receive a paper questionnaire during the month following COVID19 related confinement and all the material to send it back to the institution. They receive the same questionnaire 3 months later with all the material to send it back to the institution. The intervention is the same for all patients wether their treatment was modified or not.

SUMMARY:
To limit Corona virus dissemination on its territory, France applied strict confinement from March 16th to May 11th. Scientific societies recommended treatment modifications and remote consultations that were applied. This study evaluates the clinical impact of these care adaptation on patients under treatment for a digestive tumor. A special focus is made on quality of life and psycho-social impact of treatment modifications on patients diagnosed with metastatic colorectal cancer and metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven digestive tumor
* Ongoing treatment from March,1st and April 30th

Exclusion Criteria:

* Patient refusal for enrollment in the study
* Patient not recognised legally competent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under chemotherapy, immunotherapy or targeted therapy for a digestive tumor had their treatment modified during Coronavirus epidemia in France.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Overall survival of patients with metastatic colorectal cancer or metastatic pancreatic cancer | 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - MOULIN Valérie, La Rochelle
  - BOURGEOIS Hugues, Le Mans
  - RANDRIAN Violaine, Poitiers

REFERENCES:
- [Derived] Randrian V, Dhimene A, Pillet A, Evrard C, Elfadel R, Boyer C, Guyot d'Asnieres de Salins A, Ingrand I, Ferru A, Rouleau L, Tougeron D. COVID-19 lockdown-related treatment modifications did not impact the outcome of digestive cancers: the Clin-COVIDICA prospective study. BMC Cancer. 2025 Mar 5;25(1):398. doi: 10.1186/s12885-025-13787-9. PMID 40045328